CLINICAL TRIAL: NCT03038165
Title: Hemodynamic Parameters Changes in the Course of Hemodialysis Sessions in Patients With Intradialytic Hypertension
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Khaled Khazim, MD, Principle investigator, Western Galilee Hospital-Nahariya
Other Study IDs: GMC170114CTIL
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Intradialytic Hypertension
Keywords: Hemodialysis; Intradialytic hypertension; Hemodynamics changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While the exact pathogenesis of Intradialytic hypertension remains to be determined, several mechanisms were proposed to be involved. The main factors to determine the arterial blood pressure are the peripheral vascular resistance and cardiac output. The assumption is that the increase of blood pressure is related to the increase in peripheral vascular resistance during the dialysis session, due to fluid removal and fast reduction of the intravascular volume reduction.

Using the NICAS device (Non-Invasive Cardiac System), the hemodynamic profile in patients with intradialytic hypertension will be evaluated

DETAILED DESCRIPTION:
The number of patients with end stage renal disease (ESRD) is growing worldwide and nowadays hemodialysis (HD) treatment is the prevalent modality of renal replacement therapy. Paradoxically an increase of BP during or immediately after the HD sessions has been observed in some patients. This phenomenon is referred to as Intradialytic Hypertension (IDH). The focus will be on systolic BP increase ≥ 10 mmHg during or immediately after hemodialysis which results in post-dialysis hypertension BP above ≥130/80 mmHg. IDH affects up to 10-15% of hemodialysis patients. Patients with IDH have unfavorable outcomes; previous epidemiological data showed that IDH is associated with higher cardiovascular morbidity and mortality rates.

From the view of hemodynamic profile, peripheral resistance and cardiac output are the most important factors contributing to arterial blood pressure. The pathogenesis of IDH is likely to be multifactorial. Several mechanisms were proposed to be involved in the pathogenesis of this phenomenon.

Endothelial dysfunction, increased activity of the renin angiotensin aldosterone system (RAAS) and activation of the sympathetic nervous system had been shown to be involved in the increase of blood pressure during Hemodialysis in this group of patients.

None of these possible explanations or their inter-relationships has been studied in a controlled experimental setting and the actual physiological changes during hemodialysis in intradialytic hypertensive patients still remain unexplored.

The NICAS (Non-Invasive Cardiac System) device, used mainly for noninvasive cardiac diagnostic purposes, is substantially equivalent to the use of other hemodynamic evaluation tools, yet it is non-invasive and provides on-line data regarding the hemodynamic status of patients. Using this device, the hemodynamic changes during the HD session of IDH patients will be investigated.

By using the NICAS device, the hemodynamics parameters changes during the dialysis session will be measured. The parameters that will be measured are heart rate, stroke volume, cardiac index, cardiac power index and total peripheral vascular resistance.

During the hemodialysis treatment several hemodynamic changes may occur due to intravascular volume reduction. Changes in peripheral vascular resistance, cardiac output and cardiac power index contribute to the hemodynamic stability during the dialysis session.

By using a non-invasive technique, the NICAS device,hemodynamic changes that occur during the hemodialysis session will be evaluated.

An increase of blood pressure is correlated with the increase of peripheral vascular resistance and/or the increase of cardiac output, reflecting an adjustment to the fast changes in the intravascular volume.

Aim of the study The hemodynamic changes that occur during the dialysis session in patients with intradialytic hypertension by using the NICAS device will be evaluated.

Methods This will be an observational prospective study that examines hemodynamic parameters before and immediately after the dialysis session.

The hemodynamic data is collected by the investigators during the study period. These parameters will be obtained before starting the dialysis session, every hour during the dialysis session and at the end of it.

ELIGIBILITY:
Inclusion Criteria:

* Intradialytic hypertension at least once weakly
* Age older than 18 years
* Chronic hemodialysis treatment more than 3 months
* Stable dialysis treatment conditions
* Stable antihypertensive treatment for the last 4 weeks prior the study
* Patients able and agree to sign the consent form.

Exclusion Criteria:

* Recent changes in the antihypertensive treatment
* Recent acute cardiovascular event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty two patients on Chronic Hemodialysis treatment that exhibit intradialytic hypertension in the dialysis unit in the Galilee Medical Center will be included during 2016-2017.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Peripheral vascular resistance (dyne/sec/cm5) | During 3 consecutive hemodialysis session in one week
  In patients with intradialytic hypertension
Stroke volume (ml) | During 3 consecutive hemodialysis session in one week
  In patients with intradialytic hypertension
Stroke index (ml/m2) | During 3 consecutive hemodialysis session in one week
  In patients with intradialytic hypertension
Cardiac output (l/min) | During 3 consecutive hemodialysis session in one week
  In patients with intradialytic hypertension
Cardiac index (l/min/m2) | During 3 consecutive hemodialysis session in one week
  In patients with intradialytic hypertension
Heart rate (bpm) | During 3 consecutive hemodialysis session in one week
  In patients with intradialytic hypertension
blood pressure (mm/Hg) | During 3 consecutive hemodialysis session in one week
  In patients with intradialytic hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No